CLINICAL TRIAL: NCT05396625
Title: Optimizing Prevention Approaches for Children Reintegrating From Orphanages in Azerbaijan
Brief Title: Reintegration of Children From Institutions in Azerbaijan
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Mental Health Centre (Unknown); SOS Children's Villages (Other); Research and Education Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB20-1018; R01HD099847 (NIH)
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Emotional Trauma; Child Mental Disorder; Child Maltreatment
Keywords: Azerbaijan; Children; Child Mental Health; Family Strengthening; Economic Empowerment; Child and Family Well-being; Child Separation; Child Maltreatment
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Schools; Referral and Consultation

STUDY DESIGN:
Intervention Model Description: The study will use a randomized design and apply MOST approach to test and compare the three intervention components: a) a family-strengthening intervention; b) mental health screening and referral for treatment; and c) economic empowerment in the form of Child Savings Accounts.
  There are three factors (intervention components) and each factor has two levels. This is a 2*2*2, or 2 by 3, factorial design and, therefore, the study will have eight different experimental conditions or groups (2 by 3=8). The eligible and consenting child-parent dyads (N=400) will be randomly assigned to one of eight study groups (50 dyads per group), determining how many and which intervention components participants will receive. Given this design, half of the sample (n=200) will receive each intervention component (e.g., families assigned to Groups 1-4 will receive the family strengthening intervention and will be compared to families from Groups 5-8). All participants will receive Usual Care.
Who Masked: Outcomes Assessor
Masking Description: The eligible and consenting child-caregiver dyads will be randomized into one of eight experimental conditions. The randomization will be performed by the Project Director immediately following the baseline visit. A secure, web-based, password-protected database built on a REDCap (Research Electronic Data Capture) platform will be used to randomize participants into the 8 experimental conditions and to manage recruitment; eligibility assessment; scheduling and tracking of baseline and follow-up assessments; and sending intervention reminders. All data collectors (or interviewers) will receive a highly structured and intensive interview training conducted by the PIs. Data collectors and outcome assessors will be masked to participants' intervention group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Family Strengthening, Mental Health, Economic Empowerment (Experimental): Group will receive: 1) Usual Care, 2) Family Strengthening, 3) Mental Health Screening & Referral, and 4) Economic Empowerment Interventions
  Interventions: Behavioral: Usual Care; Behavioral: Family Strengthening; Behavioral: Mental Health Screening, Referral and Connection to Services; Other: Economic Empowerment
- Family Strengthening, Mental Health (Experimental): Group will receive: 1) Usual Care, 2) Family Strengthening, and 3) Mental Health Screening & Referral Interventions
  Interventions: Behavioral: Usual Care; Behavioral: Family Strengthening; Behavioral: Mental Health Screening, Referral and Connection to Services
- Family Strengthening, Economic Empowerment (Experimental): Group will receive: 1) Usual Care, 2) Family Strengthening, and 3) Economic Empowerment Interventions
  Interventions: Behavioral: Usual Care; Behavioral: Family Strengthening; Other: Economic Empowerment
- Family Strengthening Only (Experimental): Group will receive: 1) Usual Care and 2) Family Strengthening Interventions
  Interventions: Behavioral: Usual Care; Behavioral: Family Strengthening
- Mental Health, Economic Empowerment (Experimental): Group will receive: 1) Usual Care, 2) Mental Health Screening & Referral, and 3) Economic Empowerment Interventions
  Interventions: Behavioral: Usual Care; Behavioral: Mental Health Screening, Referral and Connection to Services; Other: Economic Empowerment
- Mental Health Only (Experimental): Group will receive: 1) Usual Care and 2) Mental Health Screening & Referral Interventions
  Interventions: Behavioral: Usual Care; Behavioral: Mental Health Screening, Referral and Connection to Services
- Economic Empowerment Only (Experimental): Group will receive: 1) Usual Care and 2) Economic Empowerment Interventions
  Interventions: Behavioral: Usual Care; Other: Economic Empowerment
- Usual Care Only (Experimental): Group will receive: Usual Care Intervention only
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Usual Care — All participants will receive the following services: case management and psychosocial support (e.g., assessment and identification of families eligible for reunification; preparing children and parents for reunification; and assistance with receiving social benefits such as Targeted Social Assistance, alimonies, or disability benefits); referrals to schools outside of their orphanage; and leisure activities for children (e.g., music, sport, and drama) provided by the orphanage staff and municipal social services.
Behavioral: Family Strengthening — Due to its focus on family-strengthening, the study uses the evidence-based intervention, SAFE Children, which employs a multiple family group format and is designed to improve family functioning, strengthen child-parent relationships and communication, enhance supportive parenting strategies, and prevent emotional and behavioral problems among at-risk children. The family-focused intervention consists of weekly multiple family group meetings (e.g. about 5 families per group). All interested family members are invited to join the sessions. The adapted intervention incorporates new sessions that address unique issues faced by families reuniting with formerly institutionalized children, such as, separation and attachment issues, children's feelings of resentment, parents' feelings of guilt and shame, stigmatized status in the community. Each session lasts about one to one and a half hours and delivered by facilitator and co-facilitator at the SOS Child and Family Center.
  Other Names: Schools and Families Educating Children
  Arms: Family Strengthening Only; Family Strengthening, Economic Empowerment; Family Strengthening, Mental Health; Family Strengthening, Mental Health, Economic Empowerment
Behavioral: Mental Health Screening, Referral and Connection to Services — Children assigned to this intervention will receive clinical assessment performed by psychiatrists at the National Mental Health Centre in Azerbaijan. From there, each child will have an individual plan developed by the multidisciplinary team and will be connected to the National Mental Health Centre clinicians to receive corresponding mental health services.
  Arms: Family Strengthening, Mental Health; Family Strengthening, Mental Health, Economic Empowerment; Mental Health Only; Mental Health, Economic Empowerment
Other: Economic Empowerment — The economic component will be in the form of Child Development Accounts/CDAs, an asset-based strategy encouraging savings and investment. This component will connect families to a bank and train them on how to save small amounts, which will be matched by contributions from the project. Matched savings will be deposited in a separate account and can be used only towards a child's education or for housing. The project will provide $50 as seed money to open a savings account in the child's name. The child's family members will make small monthly contributions to the CDA, and savings of up to $20 per month will be matched with project funds at a rate of 2:1. Caregivers will also receive training on savings and financial planning. The curriculum will be taught by trainers from the SOS in a group format for 5 sessions and will cover these topics: The Importance of Saving; Identifying and Managing Resources; Setting Up a Savings System; Sources of Income; and Budgeting and Spending.
  Arms: Economic Empowerment Only; Family Strengthening, Economic Empowerment; Family Strengthening, Mental Health, Economic Empowerment; Mental Health, Economic Empowerment

SUMMARY:
To prevent mental health problems among 7-12 children from orphanages reunited with their biological or extended families in Azerbaijan, this study will refine and test three evidence-based intervention approaches (a) family strengthening intervention; b) mental health screening and referral for treatment; and c) economic empowerment in the form of Child Development Accounts.

The study will use a randomized experimental design and participating families will be assigned to receive the family strengthening, mental health, or economic interventions. Eligible and consenting 400 child-caregivers dyads will complete baseline, 1-year, and 2-year follow-up measures. Additionally, post-intervention qualitative interviews (n=60) will solicit narrative information about participants' and services providers' reactions and experiences with each intervention component and will provide more comprehensive evidence about the interventions' efficacy.

It is hypothesized that by enhancing children's coping skills, strengthening child-parent relationships, and reducing parental stress, an intervention can help children demonstrate fewer symptoms of: a) disturbances of attachment; b) internalizing problems (depressive or anxious mood), c) externalizing problems (aggressive, delinquent, or disruptive behaviors); d) post-traumatic stress; and e) lower prevalence of diagnoses (e.g. depression, anxiety, PTSD, oppositional-defiant disorder, and reactive attachment disorder).

DETAILED DESCRIPTION:
The countries of the former Soviet Union (fSU) and Eastern Europe have the highest number of children in institutional care worldwide--up to 1.3 million children. Institutional care is associated with severe developmental setbacks and poor mental health outcomes for children, and many fSU countries are looking to develop reintegration programs supported by evidence.

Acknowledging the detrimental effects of institutionalization on children, the government of Azerbaijan jointly with UNICEF is implementing a national de-institutionalization program (De-I) aiming to close down orphanages and place children in family-oriented care. The De-I program provides basic case management services to reunite children with their families of origin, but does not address mental health needs of institutionalized children, who after years of isolation, maltreatment and traumatic experiences in orphanages, are returning home to parents who are unprepared to deal with the emotional and behavioral problems of their children. In addition, the current De-I model does not address the family-level poverty which led to institutionalization in the first place, creating a risk for future abandonment and poor psychosocial outcomes.

This study focuses on building research capacity in the field of global mental health to identify effective prevention strategies and develop innovative psychosocial intervention models tailored to the local context of post-Soviet countries. According to the National Institute of Mental Health Grand Challenges in Global Mental Health, advancement of prevention and implementation of early interventions (Goal B) is among the key global mental health priorities. Early prevention reduces the risk of developing mental disorders in adulthood, has long-term impact and may concurrently affect a number of psychosocial outcomes. There are no evidence-based, culturally-tailored, preventive mental health interventions available for institutionalized children in Azerbaijan and other fSU countries. Existing interventions in the U.S. often require highly skilled clinicians and are not adapted for the context of developing countries with limited financial and human mental health resources.

Effective parenting and behavior management skills are essential for preventing emotional and behavioral problems among children. However, in low-resource settings, non-parenting factors such as poverty induced parental stress have also been linked to poor child mental health outcomes and cannot be addressed by parenting skills programs alone. Based on the formative research conducted by the investigative team (2014-2018) in collaboration with a local Community Collaborative Board (CCB), we selected and adapted empirically-tested intervention components to ensure their cultural relevance, viability and inexpensive delivery, essential for developing countries. To promote family stability and improve the emotional well-being among children reuniting with psychosocial functioning of institutionalized children, the proposed intervention will include three components: a) a family-strengthening program, b) referral and access to mental health treatment; and c) economic empowerment. The proposed study will test these intervention components with 400 child-parent dyads in a trial using the Multiphase Optimization Strategy (MOST) to compare different intervention components and identify the most optimal combination. If efficacious, the optimized intervention may enhance the traditional De-I model and be scaled up throughout Azerbaijan and other fSU countries.

The specific aims of the research study within the R01 mechanism are:

Aim 1: To refine, test and compare the effects of three intervention components (family strengthening intervention; referral and access to mental health treatment; and economic empowerment) on mental health outcomes (a) post-traumatic symptoms; b) disturbances of attachment; c) internalizing problems--depression, anxiety; and d) externalizing problems--aggressive or disruptive behavior) among 7-12 year old children from orphanages re-entering family contexts in Azerbaijan.

Aim 2: To examine the role of hypothesized intervention mediators (emotion regulation, supportive parenting, and parental stress) and moderators (child's age, gender, length in institution, family structure, and intervention adherence) in improvements in child mental health outcomes.

Aim 3: To explore facilitating factors and barriers to implementation and participation in each intervention component (at individual, family, and organizational levels) using qualitative interviews with intervention participants and service providers. We will also conduct a secondary analysis to estimate the preliminary costs (operations and personnel) of each intervention component compared to the usual care alone.

ELIGIBILITY:
Inclusion Criteria:

1. The child is between ages 7 and 12;
2. The caregiver is at least 18 years old;
3. The child has a history of institutionalization (lived in an orphanage or another institution in Azerbaijan for a minimum of one month);
4. The child has been reunited with a caregiver (biological parent or kin relative) within a year prior to the study;
5. The child has a caregiver who is a biological parent or kin relative (e.g., grandparent) who serves as the primary caregiver;
6. The child and caregiver can commit to study participation.

Exclusion Criteria:

1. Child is not between the ages of 7-12.
2. Caregiver is below the age of 18.
3. Eligible child and/or caregiver cannot commit to study participation.
4. Children or caregivers with significant cognitive, behavioral, and/ or mental health impairment (e.g., severe developmental disorder, psychosis, severe symptoms of trauma) that may interfere with their ability to consent to and/or benefit from the program or to participate safely will also be excluded from the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in child mental health measured using the Strengths and Difficulties Questionnaire (SDQ) | Baseline, 12 months, 24 months
  Questions assess child's internalizing problems (depression, anxiety) and externalizing problems (aggressive or disruptive behavior). SDQ includes five scales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behaviors reported by parent/caregiver and teacher. With the exception of prosocial behaviors, lower score indicates reduction in mental health symptoms.
Changes in child self-reported symptoms of depression using the Center for Epidemiological Studies Depression Scale for Children (CES-DC) | Baseline, 12 months, 24 months
  The Center for Epidemiological Studies Depression Scale for Children (CES-DC) is a 20 item self-report questionnaire for young people between the ages of 6 and 17. Possible scores ranging from 0 to 60 and lower score indicates a reduction in depressive symptoms.
Changes in child's post-traumatic symptoms using the Revised Child Impact of Events Scale | Baseline, 12 months, 24 months
  Revised Child Impact of Events Scale (CRIES-8) is a 8-item child-friendly measure designed to screen children at risk for Post-Traumatic Stress Disorder (PTSD). the CRIES-8 has two sub-scales (Intrusion and Avoidance). Total scores range from 0 to 40, with higher scores indicated higher PTSD symptoms. A reduction in trauma symptoms would indicate improvement.

SECONDARY OUTCOMES:
Change in supportive parenting | Baseline, 12 months, 24 months
  The use of harsh parenting practices and level of parental support using Parenting Styles & Dimensions Questionnaire - Short version (PSDQ-Short Version). The scale includes 32 items and can be grouped into three styles and seven dimensions of parenting (e.g., physical coercion, verbal hostility, and punishment; support and affection, regulation, and autonomy). The score in all dimensions and styles ranges from 1 to 5, with higher scores indicating more use of its dimensions or styles.
Change in parental stress | Baseline, 12 months, 24 months
  The parental level of distress is measured using the Depression Anxiety Stress Scale - 21 items / DASS-21). The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. The scores for each of three sub-scales range from 0 to 42. Lower DASS score would indicate a reduction in the level of stress and anxiety among parents.
Changes in savings | Baseline, 12 months, 24 months
  Monthly savings in the Child Savings Accounts are collected through participant's bank statements. Higher average monthly saving amount would indicate improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ismayilova, PhD, Principal Investigator — University of Chicago
Locations (2):
- Azerbaijan (2):
  - National Mental Health Centre under the Ministry of Health, Republic of Azerbaijan, Baku
  - Research and Education Center, Baku

IPD SHARING:
Plan to Share IPD: Yes
Datasets will be made available to any individual who makes a direct request to the PIs and indicates the data will be used for the purposes of research (per Code of Federal Regulation Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge.").
  Shared data will be free of identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of the identity of individual subjects. Data will be shared in electronic format native to the software used by the Investigators; requestors are expected to handle converting electronic formats (though the Investigators will consider converting to tab-delimited text format if possible).
Supporting Information: Study Protocol
Time Frame: Once all of the data have been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community.
  Upon completion of the deliverable(s), the requestor will be instructed to destroy all copies of the data. If deliverables have not been produced yet, the agreement to share data will be revisited annually to decide to continue sharing or terminate the sharing agreement. If the Investigators determine that the sharing agreement should be terminated, the requestor will be instructed to destroy all copies of the data.
Access Criteria: The University of Chicago has a data sharing agreement that specifies the following conditions be met before data are shared:
  1. A formal research question is specified a priori;
  2. Names, affiliations, and roles of any other individuals who will access the shared data;
  3. The deliverable(s)-e.g., manuscript, conference presentation-are specified a priori;
  4. Proper credit and attribution-e.g., authorship, co-authorship, and order-for each deliverable are specified a priori;
  5. A statement indicating an understanding that the data can not be further shared with any additional individual(s) or parties without the PI's permission;
  6. Institutional Review Board approval for use of the data (or documentation that Institutional Review Board has determined the research is exempt);